CLINICAL TRIAL: NCT03786211
Title: The Success of the Inferior Alveolar Nerve Block Anesthesia With Alveolar Nerve Localization by Using of Panoramic Radiography in Comparison to Routine IAN Block Anesthesia: RCT
Brief Title: IANB Success Rate With and Without Panoramic Help
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hormozgan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Sajad Ansari Fard, PhD, Student research committee, Hormozgan University of Medical Sciences
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: HMS 50126
Record Dates: First submitted 2018-12-08; First posted 2018-12-24 (Actual); Last update posted 2018-12-24 (Actual); Status verified 2018-12

CONDITIONS: Anesthesia; Anesthesia; Functional
Keywords: Mandible; Anesthesia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IANB without panoramic (Active Comparator): They will get Ianb without using panoramic
  Interventions: Procedure: IANB by the guide of Panoramic; Procedure: IANB without the guide of Panoramic
- IANB with panoramic (Experimental): They will get IANB by the guide of panoramic
  Interventions: Procedure: IANB by the guide of Panoramic; Procedure: IANB without the guide of Panoramic

INTERVENTIONS:
Procedure: IANB by the guide of Panoramic — IANB will be injected by the guide of panoramic radiograph
Procedure: IANB without the guide of Panoramic — IANB will be injected without the guide of panoramic radiograph, in the routine way.

SUMMARY:
Since it is difficult to achieve anesthesia in lower jaw and the success rate of IANB is low and there are a lot of anatomic variations for the location of inferior alveolar nerve in different races, investigators decided to compare the success rate of inferior alveolar nerve block, with and without using a panoramic radiograph in Bandar Abbas population, and see if using a panoramic radiograph can increase the preciseness of the injection.

DETAILED DESCRIPTION:
This is a double blinded cross-over randomized controlled trial study conducted on all the patients of the dental clinic indicated for bilateral extraction or filling.

The randomization method is block balanced randomization. All patients will ask to fulfill the ethical Form. This form acquired demographic information (e.g. age, sex) about patients. A panoramic radiograph will take from those who matched the inclusion criteria and signed the agreement. Then a tooth from one side will be treated and the tooth from the other side of the mouth will treat at least 2 weeks later by the same dentist.

ELIGIBILITY:
Inclusion Criteria:

* Patients indicated for bilateral tooth extractions of fillings.
* Physically and mentally healthy patients who could express their pain.
* having panoramic radiograph from the past six months for other dental purposes.

Exclusion Criteria:

* sensitive to the regular anesthetics containing epinephrine.
* patients with acute or chronic pericoronitis.
* pregnancy
* trismus

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-11-12 (Actual); Primary Completion 2019-01 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Number of participants with good Anesthesia | 30 minutes after injection

CONTACTS AND LOCATIONS:
Overall Officials: Hossein Dabbagh, Md, PhD, Study Chair — Persian Gulf Oral and Dental Diseases Research Center, Hormozgan University of Medical Sciences, Bandar Abbas, Iran.
Locations (1):
- Dental clinic of BandarAbbas faculty of dentistry, BandarAbbas, Hormozgan, Iran

IPD SHARING:
Plan to Share IPD: Yes